CLINICAL TRIAL: NCT04312841
Title: Letermovir for Cytomegalovirus Prophylaxis in Patients With Hematological Malignancies Treated With Alemtuzumab
Brief Title: Letermovir for the Prevention of Cytomegalovirus Reactivation in Patients With Hematological Malignancies Treated With Alemtuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, John Reneau, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19289; NCI-2020-00169 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: B-Cell Prolymphocytic Leukemia; Chronic Lymphocytic Leukemia; Peripheral T-Cell Lymphoma; Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Sezary Syndrome; T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Leukemia, Prolymphocytic, T-Cell | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (letermovir) (Experimental): Beginning within 7 days of the first administration of standard alemtuzumab, patients receive letermovir PO (or IV over 1 hour if patient is unable to take PO for an extended period of time) daily on days 1-28. Cycles repeat every 28 days for up to 3 months after the last dose of alemtuzumab in the absence of unacceptable toxicity.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Given PO
  Other Names: 2-((4S)-8-Fluoro-2-(4-(3-methoxyphenyl)piperazin-1-yl)-3-(2-methoxy-5-(trifluoromethyl)phenyl)-4H-quinazolin-4-yl)acetic Acid; AIC246; MK-8228; Prevymis

SUMMARY:
This phase II trial studies how well letermovir works for the prevention of cytomegalovirus reactivation in patients with hematological malignancies treated with alemtuzumab. Patients receiving treatment with alemtuzumab may experience cytomegalovirus reactivation. Letermovir may block cytomegalovirus replication and prevent infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the rate of cytomegalovirus (CMV) reactivation in patients treated with letermovir at 3 months after completion of alemtuzumab therapy.

SECONDARY OBJECTIVES:

I. To evaluate the tolerability of letermovir in combination with alemtuzumab.

II. To evaluate the efficacy of letermovir for the prevention of clinically significant CMV disease.

III. To estimate the progression free survival of patients in the study population.

IV. To estimate the overall survival of patients in the study population.

EXPLORATORY OBJECTIVE:

I. To evaluate mechanisms of antiviral resistance in letermovir prophylaxis failures.

OUTLINE:

Beginning within 7 days of the first administration of standard alemtuzumab, patients receive letermovir orally (PO) (or intravenously [IV] over 1 hour if patient is unable to take PO for an extended period of time) daily on days 1-28. Cycles repeat every 28 days for up to 3 months after the last dose of alemtuzumab in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T-cell or B-cell prolymphocytic leukemia, chronic lymphocytic leukemia, peripheral T-cell lymphoma, cutaneous T-cell lymphoma, or Sezary syndrome
* Intent to treat with alemtuzumab. Monotherapy or combination with chemotherapy is allowed
* Confirmed seropositivity for CMV IgG (>= 0.7 U/mL) within 1 year of first letermovir dose
* Confirmed lack of active CMV infection as evidenced by:

  * Undetectable CMV deoxyribonucleic acid (DNA) by Abbott RealTime CMV in vitro polymerase chain reaction assay (< 50 IU/mL) within 7 days of first letermovir dose AND
  * Negative CMV IgM (< 30 AU/mL) within 7 days of first letermovir dose
* Able to provide informed consent
* Life expectancy > 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Highly unlikely to become pregnant or impregnate a partner by meeting at least one of the following:

  * A female subject who is not of reproductive potential is eligible without requiring the use of contraception. A female subject who is not of reproductive potential is defined as one who:

    * Has reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone [FSH] levels in the postmenopausal range as determined by the local laboratory, or 12 months of spontaneous amenorrhea) OR
    * Is 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy OR
    * Has undergone bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes amenorrhea (e.g., anorexia nervosa)
  * A male subject who is not of reproductive potential is eligible without requiring the use of contraception. A male subject who is not of reproductive potential is defined as one whom has undergone a successful defined as:

    * Microscopic documentation of azoospermia OR
    * A vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy
  * A male or female subject who is of reproductive potential agrees to true abstinence or to use (or have their partner use) an acceptable method of birth control starting from the time of consent through 90 days after the last dose of study therapy. True abstinence is defined as abstinence in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., abstinence only on certain calendar days, abstinence only during ovulation period, use of symptothermal method, use of post-ovulation methods) and withdrawal are not acceptable methods of contraception. Acceptable methods of birth control are:

    * Intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, and vasectomy OR use of appropriate double barrier contraception. Hormonal contraceptives (e.g., birth control pills, transdermal patch, or injectables) are also acceptable

Exclusion Criteria:

* History of confirmed CMV disease within 1 year of study entry
* History of prior allogeneic hematopoietic stem cell transplant
* End stage renal disease with creatinine clearance < 10 mL/min as defined by Cockcroft-Gault equation using serum creatinine within 7 days of enrollment
* Child-Pugh class C within 7 days of enrollment
* Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN

  * Note: Subjects who meet this exclusion criterion may, at the discretion of the investigator, have one repeat testing done. If the repeat value does not meet this criterion, they may continue in the screening process. Only the specific out of range value should be repeated (not the entire panel)
* Both moderate hepatic insufficiency AND moderate renal insufficiency:

  * Moderate hepatic insufficiency is defined as Child Pugh Class B
  * Moderate renal insufficiency is defined as a creatinine clearance less than 50 mL/min, as calculated by the Cockcroft-Gault equation
* Cytopenias are NOT an exclusion criteria in this trial as cytopenias are common in this patient population and letermovir has no known adverse effects on blood counts. Patients will be treated per institutional standard of care with as needed transfusions and growth factor support
* Received any of the following drugs within 7 days of enrollment or plans to receive any of the following during the study:

  * Ganciclovir
  * Valganciclovir
  * Foscarnet
  * Acyclovir (at doses > 3200 mg PO per day or > 25 mg/kg IV per day)
  * Valacyclovir (at doses > 3000 mg PO per day)
  * Famciclovir (at doses > 1500 mg PO per day)
  * Cyclosporine A
  * Pimozide
  * Ergot alkaloids (ergotamine and dihydroergotamine)
  * Atorvastatin at doses greater than 20 mg daily
* Received any of the following within 30 days prior to enrollment

  * Cidofovir
  * CMV hyper-immune globulin
  * Any investigational CMV antiviral agent/biologic therapy
* Infection or underlying disease necessitating ongoing use of prohibited medications
* Suspected or known hypersensitivity to active or inactive ingredients of letermovir formulations
* Positive at the time of screening for:

  * Human immunodeficiency virus (HIV) with CD4 count < 350. If HIV positive, must remain on antiretroviral therapy that is not anticipated to interact with letermovir throughout study
  * Hepatitis B surface antigen or core antibody positivity associated with detectable viral load. For any patient with serologic evidence of prior infection but undetectable viral load, viral load and surface antigen will be monitored every 2 weeks. Those with evidence of reactivation (detectable viral load) will be treated with entecavir or lamivudine. Upon resolution of detectable viral load, the patient will be allowed to continue on trial assuming adequate liver function as defined above. Alternatively, patients may be put on prophylactic entecavir or lamivudine to prevent hepatitis B reactivation at the investigator's discretion
  * Hepatitis C if no prior or current curative antiviral therapy. For those currently on curative antiviral therapy, they will be allowed on trial if hepatitis C virus (HCV) quantitation is below the limit of detection and adequate liver function as above
* Pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through 90 days after the last dose of study therapy
* Expecting to donate eggs or sperm starting from the time of consent through 90 days after the last dose of study therapy
* Currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5X half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. Subjects previously treated with a monoclonal antibody will be eligible to participate after a 28-day washout period
* Previous participation in a study using letermovir
* Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or would be put at undue risk as judged by the investigator, such that it is not in the best interest of the subject to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Reneau, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Letermovir)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 74 [56 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Performance Status [Count of Participants; unit: Participants]
  Fully Active | 2
  Restricted | 2
  Ambulatory | 1
  Unknown | 1
Histology [Count of Participants; unit: Participants]
  CTCL-Sezary Syndrome | 1
  Erythrodermic Mycosis Fungoides | 1
  T-cell Lymphoproliferative Disorder | 1
  T-cll Prolymphocytic Leukemia | 1
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Cytomegalovirus (CMV) Reactivation
Description: Defined as the proportion of patients who experience CMV reactivation (CMV deoxyribonucleic acid [DNA] by real time polymerase chain reaction > 500 IU/mL) during prophylaxis period among all patients who receive >= 90% of planned letermovir doses. The rate will be provided with 95% binomial confidence interval.
Time Frame: During prophylaxis treatment (3 months after last dose of alemtuzumab)
Population: Data for this outcome was not collected
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events Grade 3 or Above
Description: Adverse event data will be described and graded per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 guidelines. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns, especially for grade 3 or above adverse events. To assess tolerability, will also capture the proportion of patients who go off treatment due to adverse events.
Time Frame: Up to 30 days post treatment, an average of 5 months
Measure: Number; unit: participants
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 6
participants
  Platelet count decreased | 3
  Anemia | 1
  Diarrhea | 1
  White blood cell decreased | 2
  Activated partial thromboplastin time prolonged | 1
  Alkaline phosphatase increased | 1
  Lymphocyte count decreased | 1
  Neutrophil count decreased | 1
  Sinus bradycardia | 1

3. Secondary Outcome: Development of CMV Disease
Description: Clinically significant CMV reactivation be determined per the Disease Definitions Working Group of the Cytomegalovirus Drug Development Forum.
Time Frame: Up to 2 years
Population: Data for this outcome was not collected
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be estimated with the method of Kaplan-Meier (KM), where KM curves will be drawn to aid with visualization and estimates provided with 95% confidence intervals.
Time Frame: From trial enrollment to the occurrence of progression and death, assessed up to 2 years
Population: Data for this outcome was not collected
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated with the method of KM, where KM curves will be drawn to aid with visualization and estimates provided with 95% confidence intervals.
Time Frame: From trial enrollment to the occurrence of death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 6
months | 8.3 [0.4 to NA] — Due to low accrual the upper limit for the confidence interval was not able to be determined.

6. Other Pre Specified Outcome: Genotyping of Mutations in CMV Terminase Complex Genes
Description: CMV DNA sequence analysis to be performed only in subjects with CMV reactivation. Resistance to letermovir will be monitored by retrospective genotypic analysis of the CMV terminase genes in CMV DNA extracts from selected plasma samples collected at the time of diagnosed CMV reactivation. Samples will be analyzed by standard population sequencing technology through an established contract laboratory with validated protocols in place.
Time Frame: Up to 2 years
Population: Data for this outcome was not collected
Arm/Group | Treatment (Letermovir)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for patients using NCI CTCAE version 5.0 from the start of study to up to 30 days after finishing the last cycle of treatment; an average of 5 months. All-Cause Mortality was monitored/assessed up to 2 years
Arm/Group | Treatment (Letermovir)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Letermovir) (N=6)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Letermovir) (N=6)
Platelet Count Decreased (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT04312841/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT04312841/ICF_000.pdf